CLINICAL TRIAL: NCT06616987
Title: A Multicenter, Open-label, Single-arm, Clinical Trial to Evaluate the Preventive Effect of Pegylated G-CSF (PG) on Neutropenia in Patients With Metastatic Triple-negative Breast Cancer (mTNBC) Receiving Sacituzumab Govitecan (SG)
Brief Title: Prevention of Sacituzumab Govitecan-related Neutropenia in Patients With Metastatic Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yeon Hee Park (Other)
Responsible Party: Sponsor-Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-09-028
Record Dates: First submitted 2024-09-19; First posted 2024-09-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Metastatic
MeSH Terms: interventions — sacituzumab govitecan; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mTNBC patient who is administered with Sacituzumab Govitecan (Experimental): ▪ Sacituzumab Govitecan group
  - Sacituzumab Govitecan 10mg/kg IV on CnD1 and D8 + Pegfilgrastim 6mg SC QD on CnD9
  Interventions: Drug: Sacituzumab Govitecan with pegfilgrastim

INTERVENTIONS:
Drug: Sacituzumab Govitecan with pegfilgrastim — ▪ Sacituzumab Govitecan group
  - Sacituzumab Govitecan 10mg/kg IV on CnD1 and D8 + Pegfilgrastim 6mg SC QD on CnD9

SUMMARY:
Prevention of Sacituzumab Govitecan-related Neutropenia in Patients with metastatic Triple Nagative Breast Cancer who have received at least one, and no more than two, prior standard of care chemotherapy regimens

DETAILED DESCRIPTION:
▪ Sacituzumab Govitecan group

- Sacituzumab Govitecan 10mg/kg IV on CnD1 and D8 + Pegfilgrastim 6mg SC QD on CnD9

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF) prior to participation in any study-related activities.
2. Patients aged ≥19 years at the time of signing ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 12 weeks.
5. Histologically confirmed TNBC per American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria based on local testing on the most recent analyzed biopsy. Triple-negative is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PgR) and negative for human epidermal growth factor receptor 2 (HER2) (0-1+ by IHC or 2+ and negative by in situ hybridization [ISH) test].
6. Metastatic disease documented by computerized tomography (CT) scan or magnetic resonance imaging (MRI) that is not amenable to resection with curative intent.
7. Refractory to at least one, and no more than two, prior standard of care chemotherapy regimens for unresectable locally advanced or MBC. PARP inhibitor could have been counted as prior chemotherapy for purposes of study eligibility.
8. All patients must have been previously treated with taxanes regardless of disease stage (adjuvant, neoadjuvant, or advanced), unless contraindicated for a given patient.
9. Measurable or non-measurable, but evaluable disease, as per RECIST v.1.1. Patients with bone-only metastases are also eligible.
10. Brain MRI must be done for patients with suspicion of brain metastases and patient must have stable central nervous system (CNS) disease for at least 4 weeks after local therapy, without neurological symptoms, and off anticonvulsants and steroids (no more than 10mg/day prednisone or its equivalent) for at least 2 weeks before first dose of study treatment.
11. Meet the following organ function requirements:

    * Hemoglobin ≥ 9 g/dL
    * ANC ≥ 1500/mm3
    * Platelets ≥ 100,000/μL
    * Bilirubin ≤ 1.5 X IULN or ≤ 3X IULN for patients with documented Gilbert's syndrome
    * AST and ALT ≤ 2.5 X IULN or ≤ 5 X IULN if known liver metastases
    * Serum albumin > 3 g/dL
    * Creatinine clearance ≥ 60 mL/min or ≥ 30 mL/min as assessed by the Cockcroft-Gault equation
    * INR/PT and PTT or aPTT ≤ 1.5 X IULN unless patient is currently receiving therapeutic anticoagulant therapy
12. Resolution of all acute AEs of prior anti-cancer therapy to grade 1 as determined by the NCI-CTCAE v.5.0 (except for alopecia or other toxicities not considered a safety risk for the patient at investigator discretion).
13. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use institution specified method(s) of contraception during treatment with sacituzumab govitecan and for 6months after the last dose.

    * Required contraception for female of childbearing potential patients using hormonally based method, intrauterine device (IUD), bilateral tubal occlusion, female condom with spermicide should during study period and continue until 6 months after the last dose of latest administered study drug
    * Required contraception for male patients using abstinence, male condom with spermicide, vasectomy should during study period and continue until 6 months after the last dose of latest administered study drug
14. Patients must have completed all prior cancer treatments at least 2 weeks prior to 1st infusion of study drug including chemotherapy (includes also endocrine treatment), radiotherapy, and major surgery.

    * Prior anticancer biologic agent must have been completed at least 4 weeks prior to 1st infusion of study drug.

Exclusion Criteria:

1. Prior treatment with topoisomerase 1 inhibitors as a free form or as other formulations.
2. Received any prior treatment with a Trop-2-directed ADC.
3. Patients with carcinomatous meningitis.
4. Known hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances.
5. Patients positive for HIV-1 or -2 with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
6. Have active hepatitis B virus (HBV) (defined as having a positive hepatitis B surface antigen test) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

   1. Patients who test positive for hepatitis B surface antigen will be excluded.
   2. Patients who test positive for hepatitis B core antibody will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease. Patients with positive hepatitis B core antibody but negative viral load by PCR may be eligible if they are being monitored for potential viral reactivation or are willing to start or maintain antiviral treatment during study conduction (as dictated by their local and institutional standard practice or guidelines). A patient with a history of HBV infection and presence of hepatitis B surface antibody may participate in the study. In this last scenario, viral load (HBV DNA) is not mandated.
   3. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require an HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
7. Scheduled surgery during the study, other than minor surgery which would not delay study drug (eg, port insertion, tooth extraction, any procedure that requires < 1-hour general anesthesia. Procedures performed under local or intravenous (IV)/monitored sedation that lasts < 2 hours are acceptable).
8. Have an active second malignancy. Note: Patients with a history of malignancy that has been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or patients with surgically cured tumors with low risk of recurrence (eg, nonmelanoma skin cancer, histologically confirmed complete excision carcinoma in situ, or similar) are eligible.
9. Known history of clinically significant bleeding, intestinal obstruction, or gastrointestinal perforation within 6 months of study initiation.
10. Active or prior documented inflammatory bowel disease (i.e. Crohn's disease, ulcerative colitis, or a preexisting chronic condition resulting in baseline grade ≥1 diarrhea).
11. Infection requiring antibiotic use within 1 week of 1st infusion of study drug.
12. Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
13. Women who are pregnant or lactating.
14. Concomitant participation in other interventional clinical trial. Note: Patients participating in observational studies are eligible.
15. Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study
16. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of first dose of study drug.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of grade ≥3 neutropenia | At the end of Cycle 2 (each cycle is 21 days)
  Incidence of grade ≥3 neutropenia after 2 cycles of treatment

SECONDARY OUTCOMES:
Safety and tolerability of the study regimen | Up to 5 years
  Incidence of AEs
Objective Response Rate | Up to 5 years
  The percentage of complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response as assessed by investigator per RECIST v1.1
Progression Free Survival | Up to 5 years
Overall Survival | Up to 5 years
  The time until defined by date of all-cause mortality from the date of 1st infusion The time until defined by date of all-cause mortality from the date of 1st infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No